CLINICAL TRIAL: NCT02630290
Title: Addition of Dexmedetomidine to Ropivacaine-induced Supraclavicular Plexus Block, a Randomized Controlled Study
Brief Title: Addition of Dexmedetomidine to Ropivacaine-induced Supraclavicular Block (ADRIB Trial)
Acronym: ADRIB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, MD, PhD, Vice-Director in Dept Anesth & Pain, Director of Dept Pain, Principle Investigator, Professor, Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GZZD-2015008
Record Dates: First submitted 2015-12-03; First posted 2015-12-15 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Radius Fractures; Ulna Fractures; Hand Injuries; Wrist Injuries; Forearm Injuries
Keywords: Brachial plexus block; Dexmedetomidine; Ropivacaine; ultrasound-guided nerve block; supraclavicular brachial plexus block
MeSH Terms: conditions — Radius Fractures; Ulna Fractures; Hand Injuries; Wrist Injuries; Forearm Injuries | interventions — Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Placebo Comparator): After a careful aspiration, 1 to 2 mL of normal saline is injected for a distribution in and around the brachial plexus. Additional needle tip repositioning and injections may be needed when the distribution is not attained. Then the study drug (0.5% ropivacaine in a total volume of 20 mL) will be injected with additional fine adjustment of the block needle under continuous ultrasound monitoring.
  Interventions: Drug: Ropivacaine
- Ropivacaine + Dexmedetomidine (Experimental): After skin infiltration with 1-2 mL of lidocaine 2%, a 21-gauge 90-mm spinal needle will be inserted into the brachial plexus sheath using in-plane technique. After a careful aspiration, 1 to 2 mL of normal saline is injected for a distribution in and around the brachial plexus. Additional needle repositioning and injections may be needed when the distribution is not attained. Then the study drug (0.5% ropivacaine plus 30 microg dexmedetomidine in a total volume of 20 mL) will be injected with additional fine adjustment of the block needle under realtime ultrasound monitoring.
  Interventions: Drug: Ropivacaine + Dexmedetomidine

INTERVENTIONS:
Drug: Ropivacaine — Ultrasound-guided supraclavicular brachial plexus block with 0.5% ropivacaine
  Other Names: placebo
  Arms: Ropivacaine
Drug: Ropivacaine + Dexmedetomidine — Ultrasound-guided supraclavicular brachial plexus block with 0.5% ropivacaine plus low-dose (30 microg) dexmedetomidine
  Other Names: experimental
  Arms: Ropivacaine + Dexmedetomidine

SUMMARY:
Dexmedetomidine, an alpha 2-adrenoreceptor agonist, has been found to exerts an excellent influences on the filed of perineural block. It could shorten the onset time and prolong the duration of the nerve block and improved postoperative pain. However, Dexmedetomidine-induced bradycardia or hypotension has recently attracted considerable attention because of potentially grave consequences, including sinus arrest and refractory cardiogenic shock. A low dose may help minimize cardiovascular risks associated with dexmedetomidine. However, few studies have addressed the clinical effects of low-dose dexmedetomidine as an perineural adjuvant. The present study was designed to test the hypothesis that low-dose dexmedetomidine added to ropivacaine would safely enhance the duration of analgesia without adverse effects when compared with ropivacaine alone. Investigators will conduct a single-center, prospective, randomized, triple-blind, controlled trial in patients undergoing elective forearm and hand surgery under ultrasound-guided supraclavicular brachial plexus block using either ropivacaine or ropivacaine plus low-dose dexmedetomidine. The primary outcome is self-reported duration of analgesia . Secondary outcomes include onset time and duration of motor and sensory block, total postoperative analgesics, and safety assessment (adverse effects and postoperative abnormal sensation).

DETAILED DESCRIPTION:
Dexmedetomidine, an alpha 2-adrenoreceptor agonist, has been found to exerts an excellent influences on the filed of perineural block. It could shorten the onset time and prolong the duration of the nerve block and improved postoperative pain. However, Dexmedetomidine-induced bradycardia or hypotension has recently attracted considerable attention because of potentially grave consequences, including sinus arrest and refractory cardiogenic shock. Although meta-analysis showed that perineural dexmedetomidine as a local anaesthetic adjuvant for neuraxial and peripheral nerve blocks produced reversible bradycardia in only 7% of brachial plexus block patients and no effect on the incidence of hypotension, various clinical studies reported a significant decrease in heart rate. A low dose may help minimize cardiovascular risks associated with dexmedetomidine. However, few studies have addressed the clinical effects of low-dose dexmedetomidine as an perineural adjuvant. The present study was designed to test the hypothesis that low-dose dexmedetomidine, which till today has not been reported in the literature, added to ropivacaine for brachial plexus block would safely enhance the duration of analgesia without adverse effects when compared with ropivacaine alone. Investigators will conduct a single-center, prospective, randomized, triple-blind, controlled trial in patients undergoing elective forearm and hand surgery under ultrasound-guided supraclavicular brachial plexus block using either 20 mL of 0.5% ropivacaine or 0.5% ropivacaine plus 30 microg dexmedetomidine. The primary outcome is self-reported duration of analgesia . Secondary outcomes include onset time and duration of motor and sensory block, total postoperative analgesics, and safety assessment (adverse effects including cardiovascular inhibitions and postoperative abnormal sensation). Data will be collected and analyzed in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Surgery: elective forearm and hand surgery under ultrasound-guided supraclavicular brachial plexus block
* American Society of Anesthesiologist(ASA) physical status of Ⅰ to III
* Age between 18 to 60 years old

Exclusion Criteria:

* Having an ongoing another clinical trials
* Taking antihypertensive drugs such as methyldopa, clonidine and other α2 receptor agonist
* Peripheral neuropathy
* Cerebrovascular disease
* Psychiatric disease
* Coagulopathies
* Pregnant women
* Liver and kidney dysfunction
* Heart failure
* Known allergy or hypersensitive reaction to dexmedetomidine or anesthetic
* Patient refusal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | up to 24 hours postoperatively
  Postoperative pain using visual analog scale (VAS, 0-100, 0 = no pain, 100 = maximum imaginable pain) will be assessed. Duration of analgesia is defined by time between administration of block and the postoperative pain >3.

SECONDARY OUTCOMES:
Blood pressure (BP) | up to 24 hours postoperatively
  Noninvasive arterial BP is measured at the non-operated arm. episode of hypotension (30% decrease in mean BP in relation to baseline values) and hypertension (30% increase in mean BP in relation to baseline values) will be recorded.
Heart rate (HR): | up to 24 hours postoperatively
  HR, bradycardia (HR < 50 beats/min), and tachycardia (HR > 100 beats/min) will be recorded at the same time as BP recording.
Peripheral oxygen saturation (SpO2) | up to 24 hours postoperatively
  SpO2 and hypoxemia (SpO2 <90%) will be recorded at the same time as BP recording.
Sensory block of median nerve | up to 30 minutes after administration of block
  is defined by pinprick sensation using a 3-point scale (0-2, 0 = normal sensation, 1 = decreased pain sensation to pinprick, 2 = loss of pain sensation to pinprick) in the median nerve locations.
Sensory block of ulnar nerve | up to 30 minutes after administration of block
  Sensory block of ulnar nerve is defined by pinprick sensation using a 3-point scale (0-2, 0 = normal sensation, 1 = decreased pain sensation to pinprick, 2 = loss of pain sensation to pinprick) in the ulnar nerve locations.
Sensory block of radial nerve | up to 30 minutes after administration of block
  Sensory block of radial nerve is defined by pinprick sensation using a 3-point scale (0-2, 0 = normal sensation, 1 = decreased pain sensation to pinprick, 2 = loss of pain sensation to pinprick) in the radial nerve locations.
Sensory block of musculocutaneous nerve | up to 30 minutes after administration of block
  Sensory block of musculocutaneous nerve is defined by pinprick sensation using a 3-point scale (0-2, 0 = normal sensation, 1 = decreased pain sensation to pinprick, 2 = loss of pain sensation to pinprick) in the musculocutaneous nerve locations.
Motor block of median nerve | up to 30 minutes after administration of block
  Motor block of median nerve is defined by thumb and fifth finger pinch.
Motor block of ulnar nerve | up to 30 minutes after administration of block
  Motor block of ulnar nerve is defined thumb and second finger pinch.
Motor block of radial nerve | up to 30 minutes after administration of block
  Motor block of radial nerve is defined by finger abduction.
Motor block of musculocutaneous nerve | up to 30 minutes after administration of block
  Motor block of musculocutaneous nerve is defined by flexion of the elbow.
Duration of motor block | up to 24 hours postoperatively
  Duration of motor block is defined as the time interval between the administration of the block and the recovery of complete motor function of the hand and forearm assessed.
Success rate of nerve block | 30 minutes after administration of block
  A successful block is defined as surgery without patient discomfort and the need for supplementation of local infiltration or general anesthesia
Postoperative analgesic requirement | up to 24 hours postoperatively
  IV tramadol 50mg will be administered when postoperative pain >3, and be titrated up by 50 mg increments as needed for pain every 4 to 6 hours, with the maximum total dose of 250mg.
Postoperative nausea and vomiting (PONV) | up to 24 hours postoperatively
  The incidence of PONV will be recorded using a 4-point objective score (1 = no PONV;2 = mild nausea, no vomiting; 3 = excessive nausea or vomiting;4 = vomiting ≥2 times).
Abnormal sensation of brachial plexus | Day 1
  Patient's self-reported abnormal sensation of the hand and forearm.

OTHER OUTCOMES:
The block performance time | 1 day
  Time elapses from probe positioning to the end of local anesthetic injection.
The number of block performance attempts | 1 day
  Number of block performance attempts

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcai Ruan, MD, PhD, Principal Investigator — Guangzhou First People's Hospital
Locations (1):
- Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wu HH, Wang HT, Jin JJ, Cui GB, Zhou KC, Chen Y, Chen GZ, Dong YL, Wang W. Does dexmedetomidine as a neuraxial adjuvant facilitate better anesthesia and analgesia? A systematic review and meta-analysis. PLoS One. 2014 Mar 26;9(3):e93114. doi: 10.1371/journal.pone.0093114. eCollection 2014. PMID 24671181
- [Result] Marhofer D, Kettner SC, Marhofer P, Pils S, Weber M, Zeitlinger M. Dexmedetomidine as an adjuvant to ropivacaine prolongs peripheral nerve block: a volunteer study. Br J Anaesth. 2013 Mar;110(3):438-42. doi: 10.1093/bja/aes400. Epub 2012 Nov 15. PMID 23161360
- [Result] Abdallah FW, Brull R. Facilitatory effects of perineural dexmedetomidine on neuraxial and peripheral nerve block: a systematic review and meta-analysis. Br J Anaesth. 2013 Jun;110(6):915-25. doi: 10.1093/bja/aet066. Epub 2013 Apr 15. PMID 23587874
- [Result] Esmaoglu A, Yegenoglu F, Akin A, Turk CY. Dexmedetomidine added to levobupivacaine prolongs axillary brachial plexus block. Anesth Analg. 2010 Dec;111(6):1548-51. doi: 10.1213/ANE.0b013e3181fa3095. Epub 2010 Oct 1. PMID 20889939
- [Derived] Liu W, Guo J, Zheng J, Zheng B, Ruan X; Addition of Dexmedetomidine to Ropivacaine-Induced supraclavicular Block (ADRIB) investigator. Low-dose dexmedetomidine as a perineural adjuvant for postoperative analgesia: a randomized controlled trial. BMC Anesthesiol. 2022 Aug 5;22(1):249. doi: 10.1186/s12871-022-01791-6. PMID 35931989